CLINICAL TRIAL: NCT03651518
Title: Personalized Targeted Therapies in Inflammatory Complex Multi Organ Disease
Brief Title: Personalized Therapies in Inflammatory Complex Disease
Acronym: PIMOC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P160906J; 2017-000519-18 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-06-25; First posted 2018-08-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Disease; Autoimmune Diseases
Keywords: Personalized treatment; Inflammatory diseases; auto-inflammatory diseases; auto-immune diseases; Targeted treatments; skin
MeSH Terms: conditions — Autoimmune Diseases | interventions — Interleukin 1 Receptor Antagonist Protein; Adalimumab; Ustekinumab; secukinumab; tocilizumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Kineret (Experimental)
  Interventions: Drug: Kineret
- Humira (Experimental)
  Interventions: Drug: Humira
- Stelara (Experimental)
  Interventions: Drug: Stelara
- Cosentyx (Experimental)
  Interventions: Drug: Cosentyx
- Roactemra (Experimental)
  Interventions: Drug: Roactemra
- Rituximab (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Kineret — 100 mg, once/day sc 6 months
  Arms: Kineret
Drug: Humira — 40 mg/15 days sc 6 months
  Arms: Humira
Drug: Stelara — 45 mg/12 weeks sc, 6 months
  Arms: Stelara
Drug: Cosentyx — 300mg sc every week for 1 month, then 300 mg/month sc for 5 months
  Arms: Cosentyx
Drug: Roactemra — 480 mg/perf/4 weeks 6 months
  Arms: Roactemra
Drug: Rituximab — 2 sessions of 1000 mg at inclusion and 15 days after inclusion
  Arms: Rituximab

SUMMARY:
Inflammatory diseases may display atypical features making such patients impossible to classify. Management of these cases in daily practice cannot rely on the results of clinical trials nor on guidelines. DNA and RNA mapping have become major tools to understand and sometimes direct the treatment strategy in oncology. This study aims to test whether a precise analysis of molecular pathways in inflammatory, non classified diseases, can constitute a predictive tool of therapeutic efficiency

DETAILED DESCRIPTION:
This is a phase IIb study. The main objective of this study is to evaluate the efficacy of targeted treatments in patients displaying a non-classified, severe and resistant inflammatory disease. Targeted treatments for each patient will have been selected through an algorithm based on molecular analysis of specific altered inflammatory signaling pathway.

Treatments consist in targeted therapies approved in other indications (Kineret®, Humira®, Stelara®, Cosentyx®, Roactemra® and Rituximab®) that will be given once selected using molecular analysis and decision making procedure by the Scientific committee.

For each patient, one targeted treatment will be administered according to the SmPC procedure for a treatment period of 6 months.

Primary efficacy endpoint:

Response will be assessed at month 6 with a composite endpoint defined as improvement of at least 2 of the 3 following parameters:

* 50% improvement of the systemic activity assessed by the clinician following a visual analog scale (0-10 mm),
* and/or 50% improvement of cutaneous activity assessed by the involved skin surface area,
* and/or 50% decrease or normalisation of biological markers of inflammation (either CRP, ESR or fibrin).

An independent adjudication committee blinded to the treatment received, will review primary endpoint for all patients based on clinical files and standardized photographs, to validate the response.

Other secondary criteria will be assessed. Overall, this study will require a molecular analysis done on patient's tissue, the final aim being to evaluate efficiency and tolerance of targeted treatments chosen in a personalized analysis when classification is impossible.

ELIGIBILITY:
Inclusion Criteria:

* Patients (men or women) aged 18 years old and over
* Patients presenting inflammatory non classified disease targeting at least 2 organs involvement: skin, lymph nodes, hemopoietic system, joints, digestive tract, eye, nerves and brain tissues, respiratory tract, cardio-vascular disorders, genito-urinary tract including kidney, musculo-skeletal tissues. Skin involvement is mandatory in order to be able to compare involved and non-involved tissue
* Signed informed consent

The disease should be considered as non-classified despite classical and adapted investigations and evaluation through expert committee meeting.

The disease alters significantly quality of life. The impairment of quality of life will be assessed based on the investigator's assessment.

The disease has been resistant to at least two prior lines of treatment [for example : Hydroxychloroquine, Chloroquine, Colchicine, Methotrexate, Ciclosporine, Azathioprine, Mycophenolate mofetil, Disulone, Corticosteroids (prednisone, prednisolone, dexamethasone, methylprednisolone…)].

Exclusion Criteria:

* Patients presenting disease which is not featured by lesional and healthy skin areas, easy to biopsy
* Patients refusing biopsies
* Pregnancy
* Women of child-bearing potential unable to receive highly efficient contraception such as combined oral contraceptives, intra-uterine disposals, hormonal implants or the use of male condoms recommended in case of unstable or irregular partner or as a replacement method for transient unacessebility to hormonal method
* Breastfeeding
* Patients presenting disease needing urgent therapeutic measures
* Patients without health insurance or social security
* Participation in another interventional trial
* Patients under legal protection
* Patients unable to respect the wash out delay of previously taken medications before biopsy and before treatment initiation :

  * Hydroxychloroquine (wash out period = 30 days)
  * Chloroquine (wash out period = 7 days)
  * Colchicine (wash out period = 7 days)
  * Methotrexate (wash out period = 7 days)
  * Ciclosporine (wash out period = 14 days)
  * Azathioprine (wash out period = 14 days)
  * Mycophenolate mofetil (wash out period = 14 days)
  * Disulone (wash out period = 7 days)
  * Corticosteroids (=prednisone, prednisolone, dexamethasone, methylprednisolone) (wash out period = 7 days for doses greater than 5mg)
* Patients with contra-indications to treatments : Severe or active infections including tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Composite clinico-biological evaluation | 6 months
  Response will be assessed at month 6 with a composite endpoint defined as improvement of at least of 2 of the 3 following parameters:
  * 50% improvement of the systemic activity assessed by the clinician following a visual analog scale (0-10), where clinician will be asked the following question: "Please indicate, according to your clinical experience and taking into account all systemic manifestations, the level of disease activity in this patient using the following scale:"
  * and/or 50% improvement of cutaneous activity assessed by the involved skin surface area (according the rule of 9%). Standardised skin pictures will be done in order to centrally review cutaneous response.
  * and/or 50% decrease or normalisation of biological markers of inflammation (either CRP, ESR or fibrin)

SECONDARY OUTCOMES:
Number of Infections | 12 months
  to evaluate tolerance
liver cell count toxicities | 12 months
  to evaluate tolerance
kidney cell count toxicities | 12 months
  to evaluate tolerance
blood cell count toxicities | 12 months
  to evaluate tolerance
Change in Physician Global Assessment (PGA) | 1 month,
  to evaluate clinical efficiency
Change in Physician Global Assessment (PGA) | 3 months,
  to evaluate clinical efficiency
Change in Physician Global Assessment (PGA) | 6 months,
  to evaluate clinical efficiency
Change in continuous PGA | 9 months
  to evaluate clinical efficiency
Change in continuous PGA | 12 months
  to evaluate clinical efficiency
Change in British Isles Lupus Assessment Group (BILAG) | 3 months
  to evaluate clinical efficiency
Change in British Isles Lupus Assessment Group (BILAG) | 6 months
  to evaluate clinical efficiency
Change in British Isles Lupus Assessment Group (BILAG) | 9 months
  to evaluate clinical efficiency
Change in British Isles Lupus Assessment Group (BILAG) | 12 months
  to evaluate clinical efficiency
Change in Systemic Lupus Erythematosus Responder Index (SRI) | 3 months
  to evaluate clinical efficiency
Change in Systemic Lupus Erythematosus Responder Index (SRI) | 6 months
  to evaluate clinical efficiency
Change in Systemic Lupus Erythematosus Responder Index (SRI) | 9 months
  to evaluate clinical efficiency
Change in Systemic Lupus Erythematosus Responder Index (SRI) | 12 months
  to evaluate clinical efficiency
Change in Cutaneous Lupus Disease Area and Severity Index (CLASI) | 3 months
  to evaluate clinical efficiency
Change in Cutaneous Lupus Disease Area and Severity Index (CLASI) | 6 months
  to evaluate clinical efficiency
Change in Cutaneous Lupus Disease Area and Severity Index (CLASI) | 9 months
  to evaluate clinical efficiency
Change in Cutaneous Lupus Disease Area and Severity Index (CLASI) | 12 months
  to evaluate clinical efficiency
Change in 36-Item Short Form Health Survey (SF36) | 3 months
  to evaluate clinical efficiency
Change in 36-Item Short Form Health Survey (SF36) | 6 months
  to evaluate clinical efficiency
Change in 36-Item Short Form Health Survey (SF36) | 9 months
  to evaluate clinical efficiency
Change in 36-Item Short Form Health Survey (SF36) | 12 months
  to evaluate clinical efficiency
Change in CRP | 1 month
  to evaluate biological efficiency
Change in CRP | 3 months
  to evaluate biological efficiency
Change in CRP | 6 months
  to evaluate biological efficiency
Change in CRP | 9 months
  to evaluate biological efficiency
Change in CRP | 12 months
  to evaluate biological efficiency
Change in ESR (Erythrocyte sedimentation rate) | 1 month
  to evaluate biological efficiency
Change in ESR (Erythrocyte sedimentation rate) | 3 months
  to evaluate biological efficiency
Change in ESR (Erythrocyte sedimentation rate) | 6 months
  to evaluate biological efficiency
Change in ESR (Erythrocyte sedimentation rate) | 9 months
  to evaluate biological efficiency
Change in ESR (Erythrocyte sedimentation rate) | 12 months
  to evaluate biological efficiency
Change in Fibrin | 1 month,
  to evaluate biological efficiency
Change in Fibrin | 3 months
  to evaluate biological efficiency
Change in Fibrin | 6 months
  to evaluate biological efficiency
Change in Fibrin | 9 months
  to evaluate biological efficiency
Change in Fibrin | 12 months
  to evaluate biological efficiency
Decreased in serum increased cytokines, in selected RNA in peripheral blood and skin specimens | 1 month
  to evaluate targeted biological efficiency
Decreased in serum increased cytokines, in selected RNA in peripheral blood and skin specimens | 3 months
  to evaluate targeted biological efficiency
Decreased in serum increased cytokines, in selected RNA in peripheral blood and skin specimens | 6 months
  to evaluate targeted biological efficiency
Decreased in serum increased cytokines, in selected RNA in peripheral blood and skin specimens | 12 months
  to evaluate targeted biological efficiency
RNA analysis of targeted cytokines and RNA sequencing | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Selim ARACTINGI, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France